CLINICAL TRIAL: NCT03628989
Title: Evaluation of Technology-Based Distractions In Pediatric Patients During Minor Procedures
Brief Title: Technology-Based Distractions During Minor Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Samuel Rodriguez, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46917
Record Dates: First submitted 2018-07-31; First posted 2018-08-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pain; Anxiety; Procedural Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cardiac Cathertization Patients (Experimental): Participants will use technology based distraction during procedure.
  Interventions: Behavioral: Use of Virtual Technology
- Allergy Patients (Experimental): Participants will use technology based distraction during procedure
  Interventions: Behavioral: Use of Virtual Technology
- Procedure-Only Patients (No Intervention)

INTERVENTIONS:
Behavioral: Use of Virtual Technology — If parent and child consent to be in the study, the clinician will offer the use of one of the technologies: Virtual Reality (VR) headset or Augmented Reality (AR) headset. Active content includes video games, interactive avatars, and interactive experiences, while passive content includes video clips and movies. All patients will be offered the opportunity to use these technologies during their minor procedures if they meet eligibility criteria. Those who decline or who are switched over to the standard of care due to patient preference, health providers monitoring and assessment during the procedure will be noted in the database.
  Arms: Allergy Patients; Cardiac Cathertization Patients

SUMMARY:
The purpose of this study is to determine if non-invasive distracting devices (Virtual Reality headset, Augmented Reality Headset) are more effective than the standard of care (i.e., no technology-based distraction) for decreasing anxiety and pain scores in pediatric patients undergoing various minor procedures (i.e lumbar punctures and cardiac catheterization). The anticipated primary outcome will be a reduction of overall cumulative medication and secondary outcomes include but are not limited to: physician satisfaction, discharge time, pain scores, anxiety scores, and procedure time.

ELIGIBILITY:
Inclusion Criteria:

* Age 17 and under
* Able to consent or have parental consent
* Undergoing minor procedures (i.e lumbar punctures, cardiac catheterization) at Lucile Packard Children's Hospital (LPCH) or Stanford Hospital facilities

Exclusion Criteria:

* People who do not consent
* Significant Cognitive Impairment
* History of Severe Motion Sickness
* Current Nausea
* Seizures
* Visual Problems
* Non-English Speaking
* Patients who clinically unstable or requires urgent/emergent intervention
* (ASA) Physical status classification class 4 or higher
* Patient or parental preference for General Anesthesia

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Measure anxiety score | Duration of procedure (usually no more than 2-4 hours)
  Numerical anxiety scale (0-10), 0 being no anxiety and 10 being the worst imaginable anxiety

SECONDARY OUTCOMES:
Parent and Child Satisfaction Questionnaire | Duration of procedure (usually no more than 2-4 hours)
  Parent and child questionnaire with 5 questions asking the individual on a scale from 1-5 how much they agree with each statement (1=Not at all, 3=A little bit, 5=A lot). It has stamens such as "Having the technology made me feel more relaxed before my procedure" or "If I ever have procedure again, I would like to use this technology"
Virtual and Augmented Reality Feedback Survey | Duration of procedure (usually no more than 2-4 hours)
  Measure satisfaction and feedback for Virtual Reality/ Augmented Reality in regards to software and hardware for future iterations.
Asses cumulative medication dosing and the duration of procedure | Duration of procedure (usually no more than 2-4 hours)
  Measure dosing requirements for anxiolytic and/or analgesic medications for participants thought their procedure. We will then compare these doses to their own historical chart data, since many of these patents come in routinely, and use their own data for intra-reliability measures.
Evaluation of Passive vs Active Interventions | Duration of procedure (usually no more than 2-4 hours)
  There is variation in the immersive technology experiences (active vs passive content), as a part of the study the investigators also aim to evaluate the degree of cognitive load which is suitable for clinical applications during minor procedures. During the participants immersive experience in either AR or VR, there are embedded questions in the experience that can gage as to the patient's emotional status (happy, sad, mad) or VAS scales (0-10, 0=no pain, 10=worst imaginable pain) that can let the research personnel know if we need to increase the cognitive load. If patients are self-reporting higher VAS scores, or aversive emotional status (i.e mad) the cognitive load will be increased to enhance the distraction experience from the procedure.

OTHER OUTCOMES:
Fear assessment | Duration of procedure (usually no more than 2-4 hours)
  Patient's fear will be assessed through the Children's Fear Scale (CFS). Patients will be shown faces showing different levels of anxiety on a scale from 0 to 4. The left-most face (minimum value of 0) shows no anxiety at all and the right-most face shows extreme anxiety (maximum value of 4). Patients look at these faces and choose the one that shows how much anxiety was felt during procedure. This will be done only for allergy patients.
Pain Assessment | Duration of procedure (usually no more than 2-4 hours)
  Patient's pain will be assessed through the Wong-Baker FACES pain rating scale from 0 to 10. The left-most face has a value of 0 meaning no pain/doesn't hurt at all and the right-most face has a value of 10 being a lot of pain/hurts as much as you can imagine. Patients will be asked which face best describes their pain levels during the procedure. This will only be done for allergy patients.
Procedural Compliance | Duration of procedure (usually no more than 2-4 hours)
  Procedural compliance is measured through modified Induction Compliance Checklist (ICC). All behaviors observed in checklist are marked. Total score is the number of categories checked, perfect score is 0. This will only be done for allergy patients.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Caruso, MD, MEd, Principal Investigator — Stanford University; Samuel Rodriguez, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No